CLINICAL TRIAL: NCT06381492
Title: Quantifying Patellar Tendon Microstructure Using Diffusion Tensor Imaging
Brief Title: Quantifying Patellar Tendon Microstructure Using DTI
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2024-0057; 1K99AR085752-01 (NIH); A536130 (Other: UW Madison); SMPH/ORTHO&REHAB/PHYS THER (Other: UW Madison); Protocol Version 10/1/2025 (Other: UW Madison)
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Patellar Tendinopathy; Anterior Cruciate Ligament Reconstruction
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Bone-patellar tendon-bone (BPTB): This group will have patellar injury confirmed through self-reported surgical history and evidence of ipsilateral BPTB graft harvest on ultrasound.
  Interventions: Device: MRI; Device: Ultrasound (US); Device: Neuromuscular electric stimulation (NMES)
- Patellar tendinopathy group: This group will have patellar tendinopathy confirmed based on International Scientific Tendinopathy Symposium Consensus on Clinical Terminology (ICON) statement, which defines patellar tendinopathy as "persistent patellar tendon pain and loss of function related to mechanical loading." Ultrasound diagnosis must confirm alteration of tendon macrostructure.
  Interventions: Device: MRI; Device: Ultrasound (US); Device: Neuromuscular electric stimulation (NMES)
- Healthy knees: Control group of participants with healthy knees
  Interventions: Device: MRI; Device: Ultrasound (US); Device: Neuromuscular electric stimulation (NMES)

INTERVENTIONS:
Device: MRI — MRI using DTI technology
Device: Ultrasound (US) — Standard US
Device: Neuromuscular electric stimulation (NMES) — Standard NMES

SUMMARY:
The goal of this observational study is to understand how diffusion tensor imaging (DTI) relates to other traditional measures and knee function. The main question it aims to answer is:

Will regions of known patellar tendon pathology present with smaller DTI scalar parameters, shorter fiber length, and lower fiber density compared to the contralateral tendon and healthy regions in the ipsilateral tendon.

Participants will:

* undergo MRI and ultrasound imaging
* perform knee function test
* complete questionnaires

DETAILED DESCRIPTION:
Patellar tendon injuries are commonly accompanied by macrostructural alterations captured on common imaging modalities, and the extent of these alterations correlate to knee joint function. Evidence for using tendon macrostructure for diagnosis and prognosis of tendon injuries is not as clear, suggesting that these imaging modalities are not providing a complete picture of the alterations. Diffusion tensor imaging (DTI) tractography can quantify tendon microstructures that underlie the alterations in pathological tendons and shows promising results in healthy tendons. This study is the first step in evaluating whether tendon microstructure captured using DTI technology can be applied as a biomarker to optimize treatment for patellar tendon injuries.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Have patellar tendon injury as confirmed through subjective report, clinical examination, and ultrasound by an experienced physical therapist
* Patellar tendinopathy group must present with current symptoms of patellar tendinopathy
* Control group must have no history of patellar tendon injury

Exclusion Criteria:

* Participants with a history of invasive procedures other than bone-patellar tendon-bone (BPTB) autograft harvest to the patellar tendon or extensor mechanism
* Participants with history of contralateral BPTB autograft harvest, or ACLR using any other graft type
* Participants with contraindications to MRI
* Participants with contraindications to NMES

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases: Adults 18 years or older with a diagnosis of patellar tendinopathy, or with a history of anterior cruciate ligament (ACL) reconstruction using bone-patellar tendon-bone autograft.
  Controls: Adults 18 years or older without a diagnosis of patellar tendinopathy or history of ACL reconstruction using bone-patellar tendon-bone autograft
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-12-27 (Actual); Study Completion 2025-12-27 (Actual)

PRIMARY OUTCOMES:
Compare scalar parameters of known patellar tendon pathology to the contralateral tendon | Up to 2 weeks
  DTI parameters will be obtained by built-in diffusion-weighted sequences on the GE MRI machine. Regions of interest will be selected using clinical scans, and region specific DTI parameters will be compared between regions and over the repeat test sessions
Compare DTI scalar parameters of known patellar tendon pathology to the healthy regions in the ipsilateral tendon | Up to 2 weeks
  DTI parameters will be obtained by built-in diffusion-weighted sequences on the GE MRI machine. Regions of interest will be selected using clinical scans, and region specific DTI parameters will be compared between regions and over the repeat test sessions
Rank patellar tendon loads during exercise | Up to 2 weeks
  Patellar tendon loads will be obtained by tensiometer measurements during common exercises for patellar tendon rehabilitation while subject wears NMES sensors. Patellar tendon loads will be compared between regions and over the repeat test sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Heiderscheit, PT, PhD, Principal Investigator — University of Wisconsin, Madison; Daniel Cobian, DPT, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No